CLINICAL TRIAL: NCT06599749
Title: Establishment and Standardization of a Platform for In-depth Tumour Profiling (TUPRO) in Patients With Advanced and Metastatic High-Grade Adenocarcinoma of Ovarian, Tubal or Peritoneal Origin - a Prospective, Multi-centre Human Research Ordinance Research Project / Category A
Brief Title: Establishment and Standardization of a Platform for In-depth Tumour Profiling (TUPRO) in Patients With Advanced and Metastatic High-Grade Adenocarcinoma of Ovarian, Tubal or Peritoneal Origin (TUPRO-Gyn)
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02052; me18Wicki
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Adenocarcinoma of Ovary; Adenocarcinoma, Tubular; Peritoneal Cancer
Keywords: Advanced Ovarian Cancer; High-Grade Adenocarcinoma; Tubal Origin; Peritoneal Origin; Metastatic Cancer; Tumour Profiling
MeSH Terms: conditions — Adenocarcinoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Tumor tissue, blood and, if applicable, ascites fluid sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective, multi-centre, exploratory research project is the establishment of a platform for in-depth tumour profiling in patients with advanced and metastatic High-Grade Adenocarcinoma (HGAC) of ovarian, tubal or peritoneal origin.

DETAILED DESCRIPTION:
TUPRO-Gyn is part of the Tumour Profiler (TUPRO) research collaboration, which aims to help generate information about patients' individual tumour biology for patients with advanced malignancies, using innovative biotechnologies and computational analyses for in-depth molecular profiling. The TUPRO-Gyn study focuses on improving treatment for patients with advanced ovarian, tubal, or peritoneal cancer, who often face poor outcomes and limited options after initial therapy. The study aims to use advanced molecular profiling technologies to identify specific characteristics of tumors that can be targeted with personalized treatments. By building a comprehensive platform for in-depth tumor analysis, the project hopes to discover new biomarkers and support future clinical trials that match treatments to the molecular profile of individual tumors, potentially leading to better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group performance status score ≤ 2 (not bedridden for more than 50% of waking hours)
* Primary or recurrent HGAC of ovarian, tubal or peritoneal origin International Federation of Gynecology and Obstetrics (FIGO) stage III or IV
* Written informed consent according to national legal and regulatory requirements prior to any project specific procedures

Exclusion Criteria:

* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the project leader may interfere with the project or affect patient compliance
* Legal incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced and metastatic High-Grade Adenocarcinoma (HGAC) of ovarian, tubal or peritoneal origin
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Sample Processing and Report Generation (1) | Through study completion, an average of 1 year
  - Number of samples with sufficient material and quality for intended analysis.
Sample Processing and Report Generation (2) | Through study completion, an average of 1 year
  - Number of successfully processed samples per technology, with quality checks passed and interpretable results generated.
Sample Processing and Report Generation (3) | Through study completion, an average of 1 year
  - Successful data transfers into the research data management system, ensuring results are timely for inclusion in the molecular research report.
Sample Processing and Report Generation (4) | Through study completion, an average of 1 year
  - Number of molecular summary reports available for the Tumour Board.
Sample Processing and Report Generation (5) | Through study completion, an average of 1 year
  - Proportion of cases where the Tumour Board found the molecular report useful for treatment recommendations.
Sample Processing and Report Generation (6) | Through study completion, an average of 1 year
  - Proportion of cases where the treating physician found the Tumour Board's recommendation useful for treatment decisions.
Sample Processing and Report Generation (7) | Through study completion, an average of 1 year
  - Types and combinations of molecular information considered useful for treatment recommendations beyond routine diagnostics.
Classification of Proposed Treatment Options | Through study completion, an average of 1 year
  Possible treatment options are classified as follows:
  * On-label molecularly matched treatment or immunotherapy (per SwissMedic), with or without radiotherapy/chemotherapy;
  * Classical chemotherapy, with or without radiotherapy (on-label if applicable);
  * Referral to a clinical trial;
  * Off-label molecularly matched treatment or immunotherapy (per SwissMedic), with or without radiotherapy/chemotherapy;
  * Off-label treatment authorized in countries with comparable standards to SwissMedic, with or without radiotherapy/chemotherapy;
  * Best supportive care (no active anti-tumor treatment). Treatment options are discussed in an interdisciplinary Tumour Board, considering patient-centered factors like previous treatments, disease history, clinical status, and patient preferences.
Classification of Tumour Board Recommendations | Through study completion, an average of 1 year
  Grading of treatment recommendations using the European Society for Medical Oncology Scale for Clinical Actionability of Molecular Targets (ESCAT):
  I-A: Randomized trials show survival improvement with a tumor's alteration-drug match.
  I-B: Non-randomized trials show benefits in a specific tumor type. I-C: Clinical benefit seen across various tumor types or in basket trials. II-A: Retrospective studies show benefit in patients with a specific alteration vs. those without.
  II-B: Trials show better drug responsiveness, but no survival data. III-A: Benefit shown in a different tumor type; limited evidence for the patient's cancer type.
  III-B: Predicted impact similar to a studied alteration, lacking data. IV-A: Pre-clinical models show alteration affects drug sensitivity. IV-B: Actionability predicted in silico. V: Targeted therapy shows responses but no improved outcomes. X: No evidence the alteration is actionable
Time to first subsequent treatment (TTFST) | Through study completion, at least 6 month of follow up
  Time to first subsequent treatment (TTFST), incl. best supportive care
Time to first subsequent treatment (TTFST) ratio | Through study completion, at least 6 month of follow up
  Time to first subsequent treatment (TTFST) ratio (TTFST 2 / TTFST 1: TTFST 2 = TTFST on current project; TTFST 1 = TTFST on previous treatment [before entering the project])
Terminations due to toxicity | Through study completion, at least 6 month of follow up
  Frequency (proportion) of patients terminating treatment due to toxicity
Survival | Through study completion, at least 6 month of follow up
  Overall survival (OS), calculated from registration until death due to any cause
Event free survival (EFS) | Through study completion, at least 6 month of follow up
  Event free survival (EFS), defined as time to treatment failure or death
Radiological tumour response | Through study completion, at least 6 month of follow up
  Proportion of patients with a radiological tumour response (complete response (CR) / partial response (PR)) according to local standards and trial protocol (in case of referral or trial)
Quality of Life (FAC-G7) questionnaire | Every 12 weeks (+/- 2 weeks) for 6 months after last tumour sampling (day 0)
  Quality of Life assessed using the Functional Assessment of Cancer Therapy - General 7 (FACT-G7) questionnaire. The FACT-G7 uses a Likert scale, where responses range from 0 (not at all) to 4 (very much). Higher scores indicate better quality of life, while lower scores suggest more severe symptoms or a poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Wicki, Prof. Dr. med., Principal Investigator — University Hospital, Zürich
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Basel
  - Kantonsspital Baselland, Liestal
  - University Hospital Zurich, Zurich